CLINICAL TRIAL: NCT00836446
Title: Effects of Physical Activity on Cardiovascular Risk Markers in School-Aged Mexican Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Collaborators: Universidad Autonoma del Estado de Mexico (Other)
Responsible Party: Margie Balas Nakash, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 212250-02211
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Obesity; Cardiovascular Disease
Keywords: school-aged; children; obesity; cardiovascular risk; physical activity
MeSH Terms: conditions — Obesity; Cardiovascular Diseases; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): 20 min. physical activity routine
  Interventions: Other: physical activity
- Group 2 (Experimental): 40 min. aerobic physical activity routine
  Interventions: Other: physical activity

INTERVENTIONS:
Other: physical activity — physical activity routines 5 times a weeks for 12 weeks.

SUMMARY:
Childhood obesity is a public health problem; in Mexican children a high prevalence of cardiovascular risk factors are present. Physical activity has been proposed as a strategy to reduce this risk. We conducted a pre-posttest intervention study of 214 school-aged Mexican children (4th to 6th grade), to assess the effects of two physical activity routines with different duration and intensity (40 minute aerobic routine vs. 20 minute routine) on cardiovascular risk markers. Physical activity routines were assigned randomly to two public schools in Toluca, Mexico (20 min: group 1 (n= 117), 40 min: group 2 (n=97)). The routines were implemented Monday through Friday for 12 weeks. Nutrition assessment was done before and after the intervention and included anthropometric measurements (weight, height, body mass index, waist circumference and body composition), blood pressure and biochemical analysis (triglycerides, total cholesterol LDL-cholesterol, HDL-Cholesterol, glucose and insulin). Heart rate was monitored 3 times during the intervention to evaluate the routine´s intensity.

ELIGIBILITY:
Inclusion Criteria:

* All children from 4th to 6th grade, from 2 public urban schools in Toluca, Estado de México

Exclusion Criteria:

* If they have a chronic disease
* If they can not do exercise
* If they have low body mass index (BMI less than 5th percentile).
* If they miss more than 20 sessions
* If they decide that they did not want to participate any more.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of physical activity routine on cardiovascular risk markers | 3 months

SECONDARY OUTCOMES:
measure heart rate to evaluate the intensity of physical activity routines | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Otilia Perichart-Perera, M.S, RD, Study Chair — Instituto Nacional de Perinatología Isidro Espionosa de los Reyes; Felipe Vadillo-Ortega, PhD, Study Chair — Instituto Nacional de Perinatología Isidro Espionosa de los Reyes; Margie Balas-Nakash, B.S, Principal Investigator — Instituto Nacional de Perinatología Isidro Espionosa de los Reyes; Roxana Valdes-Ramos, D.Sc, Study Director — Universidad Autónoma del Estado de México. Facultad de Medicina; Alejandra D Benitez-Arciniega, M.Ph, Study Chair — Universidad Autónoma del Estado de México. Facultad de Medicina
Locations (1):
- Universidad Autonoma del Estado de Mexico, México, Toluca, Estado de Mexico, Mexico